CLINICAL TRIAL: NCT06201559
Title: An Open Label, Balanced, Randomized, Two-Treatment, Four-Period, Two-Sequence, Single Oral Dose, Full Replicate Crossover, Bioequivalence Study of Albendazole Tablets IP 400 mg of Biddle Sawyer Limited (GSK Group Company) With Albendazole Tablets 400 mg of Glaxo SmithKline Consumer Healthcare, South Africa (PTY) Ltd in Healthy, Adult Participants Under Fed Condition
Brief Title: Bioequivalence Study Between Two Albendazole 400 mg Tablets in Healthy Adult Participants Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 221030
Record Dates: First submitted 2023-12-30; First posted 2024-01-11 (Actual); Results first posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2024-12

CONDITIONS: Intestinal Diseases
Keywords: Albendazole; Bioequivalence
MeSH Terms: conditions — Intestinal Diseases | interventions — Albendazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence TRTR (Experimental): Participants will be administered with test (T) intervention [Albendazole Indian Pharmacopoeia (IP) 400 mg] in Period 1, reference (R) intervention (Albendazole Tablets 400 mg) in Period 2, T intervention in Period 3 and R intervention in Period 4.
  Interventions: Drug: Albendazole IP 400 mg
- Sequence RTRT (Experimental): Participants will be administered with reference (R) intervention in Period 1, test (T) intervention in Period 2, R intervention in Period 3 and T intervention in Period 4.
  Interventions: Drug: Albendazole 400 mg

INTERVENTIONS:
Drug: Albendazole IP 400 mg — Albendazole IP 400 mg tablets will be administered under fed conditions
  Arms: Sequence TRTR
Drug: Albendazole 400 mg — Albendazole 400 mg tablets will be administered under fed conditions
  Arms: Sequence RTRT

SUMMARY:
The goal of this study is to compare two formulations of Albendazole of the same dose in healthy adult participants. Researchers will compare the extent and rate to which the drug is absorbed.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, non-smoker, adult participants having body mass index (BMI) between 18.5 to 30.0 (both inclusive), calculated as weight in kilogram (kg)/ height in meter square (m2)
2. Not having any significant diseases or clinically significant abnormal findings during screening, medical history, clinical examination, laboratory evaluations, 12-lead electrocardiogram (ECG) and X-ray chest (postero-anterior view) recordings.
3. Able to understand and adhere to the study procedures
4. Voluntary written informed consent is given for study participation
5. In case of female participants:

Surgically sterilized at least 6 months prior to study participation;Or If of childbearing potential is willing to use a suitable and effective double barrier contraceptive method or intra uterine device during the study, And Serum pregnancy test must be negative.

Exclusion Criteria:

1. Known hypersensitivity or idiosyncratic reaction to albendazole or any excipients or any related drug or any substance.
2. History or presence of any disease or condition which might compromise the haemopoietic, renal, hepatic, endocrine, pulmonary, central nervous, cardiovascular, immunological, dermatological, gastrointestinal or any other body system.
3. Any history or presence of asthma (including aspirin induced asthma) or nasal polyp or non-steroidal anti inflammatory drugs (NSAIDs) induced urticaria.
4. History or presence of seizure or psychiatric disorders.
5. Ingestion of a medication (prescribed medication & over the counter (OTC) medication, herbal remedies, cimetidine, praziquantel, dexamethasone, ritonavir, phenytoin, carbamazepine, phenobarbital) at any time in 14 days prior to dosing and any vaccine (including COVID-19 vaccine) from 14 days prior to dosing. In any such case participant selection will be at the discretion of the Principal Investigator.
6. Receipt of an intervention or participation in a drug research study within a period of 90 days prior to the first dose of study intervention **.

   * If intervention is received within 90 days where there is no blood loss except safety lab testing, participant can be included considering 10 half-lives duration of intervention received.
7. A positive hepatitis screen including hepatitis B surface antigen and/or hepatitis C virus (HCV) antibodies.
8. A positive test result for HIV antibody (1 and/or 2).
9. The presence of clinically significant abnormal laboratory values during screening.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2023-08-21 (Actual); Primary Completion 2023-09-12 (Actual); Study Completion 2023-09-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- GSK Investigational Site, Ahmedabad, India

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/

RESULTS

PARTICIPANT FLOW:
Groups:
- Test(T) Albendazole vs Reference(R) Albendazole First,Then (T) Albendazole vs (R) Albendazole (TRTR): Participants were orally administered with Albendazole [Indian Pharmacopoeia (IP)] 400 mg (T1) tablet as single dose treatment under fed conditions on Day 1 in Period 1, followed by single dose of Albendazole 400 mg (R1) tablet in Period 2, then single dose Albendazole IP 400 mg (T2) tablet in Period 3 further followed by single dose Albendazole 400 mg (R2) tablet in Period 4
- (R) Albendazole vs (T) Albendazole First,Then (R) Albendazole vs (T) Albendazole (RTRT): Participants were orally administered with Albendazole 400 mg (R1) tablet as single dose treatment under fed conditions on Day 1 in Period 1, followed by single dose of Albendazole IP 400 mg (T1) tablet in Period 2, then single dose Albendazole 400 mg (R2) tablet in Period 3 further followed by single dose Albendazole IP 400 mg (T2) tablet in Period 4
Period: Period 1
Arm/Group | Test(T) Albendazole vs Reference(R) Albendazole First,Then (T) Albendazole vs (R) Albendazole (TRTR) | (R) Albendazole vs (T) Albendazole First,Then (R) Albendazole vs (T) Albendazole (RTRT)
Started | 35 | 35
Completed | 35 | 35
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Test(T) Albendazole vs Reference(R) Albendazole First,Then (T) Albendazole vs (R) Albendazole (TRTR) | (R) Albendazole vs (T) Albendazole First,Then (R) Albendazole vs (T) Albendazole (RTRT)
Started | 34 (One participant discontinued on own accord from Period 2 but was present in periods 3 and 4. This participant has completed the study.) | 34 (One participant withdrew from the study after completing Period 1.)
Completed | 34 | 34
Not Completed | 0 | 0
Period: Period 3
Arm/Group | Test(T) Albendazole vs Reference(R) Albendazole First,Then (T) Albendazole vs (R) Albendazole (TRTR) | (R) Albendazole vs (T) Albendazole First,Then (R) Albendazole vs (T) Albendazole (RTRT)
Started | 35 | 34
Completed | 35 | 34
Not Completed | 0 | 0
Period: Period 4
Arm/Group | Test(T) Albendazole vs Reference(R) Albendazole First,Then (T) Albendazole vs (R) Albendazole (TRTR) | (R) Albendazole vs (T) Albendazole First,Then (R) Albendazole vs (T) Albendazole (RTRT)
Started | 33 (One participant withdrew from the study after completing periods 1, 2 and 3, and another participant discontinued from Period 4 on medical ground but did not withdraw from the study.) | 32 (One participant withdrew from the study after completing periods 1, 2 and 3, and another participant discontinued on own accord from Period 4 but did not withdraw from the study.)
Completed | 33 | 32
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Test(T) Albendazole vs Reference(R) Albendazole First,Then (T) Albendazole vs (R) Albendazole (TRTR) | (R) Albendazole vs (T) Albendazole First,Then (R) Albendazole vs (T) Albendazole (RTRT) | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32 (5.25) | 34.5 (6.40) | 33.2 (5.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 31 | 31 | 62
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 35 | 35 | 70
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax) of Albendazole
Description: Blood samples were collected for pharmacokinetic (PK) analysis of Albendazole. PK parameter was determined using standard non-compartmental methods.
Time Frame: Pre-dose, 0.33, 0.67, 1, 1.33, 1.67, 2, 2.33, 2.67, 3, 3.33, 3.67, 4, 4.50, 5, 6, 8, 10, 12, 14, 18 and 24 hours
Population: PK population included all participants in Safety set who had at least 1 measurable PK assessment. As pre-specified in Statistical Analysis Plan (SAP), data is collected and reported for PK parameters per study intervention i.e. Test Study Intervention-T1 (1st administration), Test Study Intervention-T2 (2nd administration), and Reference Study Intervention-R1 and Reference Study Intervention-R2 similarly. Only those participants with data available at specified time points have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/millilitre (ng/mL)
Groups:
- Albendazole IP 400 mg/400mg - Test 1 (T1); Albendazole IP 400 mg/400 mg - Test 2 (T2); Albendazole 400 mg/IP 400 mg - Reference 1 (R1); Albendazole 400 mg/IP 400 mg - Reference 2 (R2): Participants were orally administered with Albendazole (400 mg or 400 mg IP) tablet as single dose treatment under fed conditions on Day 1 in Periods 1, 2, 3 and 4.
Arm/Group | Albendazole IP 400 mg/400mg - Test 1 (T1) | Albendazole IP 400 mg/400 mg - Test 2 (T2) | Albendazole 400 mg/IP 400 mg - Reference 1 (R1) | Albendazole 400 mg/IP 400 mg - Reference 2 (R2)
Number analyzed (Participants) | 64 | 61 | 63 | 62
nanogram/millilitre (ng/mL) | 43.846 (114.1) | 41.685 (110.9) | 39.737 (112.1) | 46.115 (102.6)
Statistical Analysis 1: Comparison: Albendazole IP 400 mg/400mg - Test 1 (T1) vs Albendazole IP 400 mg/400 mg - Test 2 (T2) vs Albendazole 400 mg/IP 400 mg - Reference 1 (R1) vs Albendazole 400 mg/IP 400 mg - Reference 2 (R2); Test type: Equivalence — Point estimate of geometric mean ratio (GMR) of T/R should be between 80.00 -125.00%. If the intra-subject variability for Cmax following replicate administrations of the comparator product was > 30%, the acceptance criteria for Cmax was widened to a maximum of 69.84-143.19%; Ratio of Geometric Least Square Means = 98.1, 90% CI 2-sided [86.79 to 110.91] — Geometric least square means were combined to perform statistical analysis of T as T1 + T2 and R as R1 + R2

2. Primary Outcome: Area Under the Plasma Concentration Curve From Time 0 to the Last Measured [AUC(0-t)] for Albendazole
Description: Blood samples were collected for PK analysis of Albendazole. PK parameter was determined using standard non-compartmental methods.
Time Frame: Pre-dose, 0.33, 0.67, 1, 1.33, 1.67, 2, 2.33, 2.67, 3, 3.33, 3.67, 4, 4.50, 5, 6, 8, 10, 12, 14, 18 and 24 hours
Population: PK population. As pre-specified in the Statistical Analysis Plan (SAP), data is collected and reported for PK parameters per study intervention i.e. Test Study Intervention-T1 (1st administration), Test Study Intervention-T2 (2nd administration), Reference Study Intervention-R1 (1st administration) and Reference Study Intervention-R2 (2nd administration). Only those participants with data available at specified time points have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour/ milliliter (ng*h/mL)
Groups:
- Albendazole IP 400 mg/400mg - Test 2 (T2); Albendazole 400 mg/ IP 400mg - Reference 1 (R1); Albendazole 400 mg/ IP 400mg - Reference 2 (R2): Participants were orally administered with Albendazole (400 mg or 400 mg IP) tablet as single dose treatment under fed conditions on Day 1 in Periods 1, 2, 3 and 4
Arm/Group | Albendazole IP 400 mg/400mg - Test 1 (T1) | Albendazole IP 400 mg/400mg - Test 2 (T2) | Albendazole 400 mg/ IP 400mg - Reference 1 (R1) | Albendazole 400 mg/ IP 400mg - Reference 2 (R2)
Number analyzed (Participants) | 63 | 60 | 63 | 62
Nanogram*hour/ milliliter (ng*h/mL) | 179.419 (129.5) | 164.052 (120.4) | 161.034 (127.4) | 182.792 (117.2)
Statistical Analysis 1: Comparison: Albendazole IP 400 mg/400mg - Test 1 (T1) vs Albendazole IP 400 mg/400mg - Test 2 (T2) vs Albendazole 400 mg/ IP 400mg - Reference 1 (R1) vs Albendazole 400 mg/ IP 400mg - Reference 2 (R2); Test type: Equivalence — Point estimate of geometric mean ratio (GMR) of T/R should be between 80.00 -125.00%. If the intra-subject variability for AUC(0-t) following replicate administrations of the comparator product was > 30%, the acceptance criteria for AUC(0-t) was widened to a maximum of 69.84-143.19%; Ratio of Geometric Least Square Means = 97.6, 90% CI 2-sided [86.86 to 109.73] — Geometric least square means were combined to perform statistical analysis of T as T1 + T2 and R as R1 + R2

3. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Albendazole Sulfoxide
Description: Blood samples were collected for PK analysis of Albendazole sulfoxide. PK parameter was determined using standard non-compartmental methods.
Time Frame: Pre-dose, 0.33, 0.67, 1, 1.33, 1.67, 2, 2.33, 2.67, 3, 3.33, 3.67, 4, 4.50, 5, 6, 8, 10, 12, 14, 18 and 24 hours
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Albendazole IP 400 mg/ 400mg - Test 1 (T1); Albendazole IP 400 mg/ 400mg - Test 2 (T2); Albendazole 400 mg/ IP 400mg - Reference 1 (R1); Albendazole 400 mg/ IP 400mg - Reference 2 (R2): Participants were orally administered with Albendazole (400 mg or 400 mg IP) tablet as single dose treatment under fed conditions on Day 1 in Periods 1, 2, 3 and 4
Arm/Group | Albendazole IP 400 mg/ 400mg - Test 1 (T1) | Albendazole IP 400 mg/ 400mg - Test 2 (T2) | Albendazole 400 mg/ IP 400mg - Reference 1 (R1) | Albendazole 400 mg/ IP 400mg - Reference 2 (R2)
Number analyzed (Participants) | 64 | 61 | 63 | 62
ng/mL | 638.051 (63.3) | 644.730 (59.4) | 643.276 (62.6) | 710.382 (53.8)

4. Secondary Outcome: Area Under the Plasma Concentration Curve From Time 0 to the Last Measured [AUC(0-t)] of Albendazole Sulfoxide
Description: as for outcome 3
Time Frame: Pre-dose, 0.33, 0.67, 1, 1.33, 1.67, 2, 2.33, 2.67, 3, 3.33, 3.67, 4, 4.50, 5, 6, 8, 10, 12, 14, 18 and 24 hours
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Albendazole IP 400 mg/ 400mg - Test 1 (T1) | Albendazole IP 400 mg/ 400mg - Test 2 (T2) | Albendazole 400 mg/ IP 400mg - Reference 1 (R1) | Albendazole 400 mg/ IP 400mg - Reference 2 (R2)
Number analyzed (Participants) | 63 | 60 | 63 | 62
ng*h/mL | 6129.744 (74.2) | 6023.449 (68.9) | 6046.054 (73.2) | 6572.338 (67.8)

5. Secondary Outcome: Area Under the Plasma Concentration-time Curve Extrapolated to Infinity [AUC0-inf] of Albendazole and Albendazole Sulfoxide
Description: Blood samples were collected for PK analysis of Albendazole and albendazole sulfoxide. PK parameter was determined using standard non-compartmental methods.
Time Frame: Pre-dose, 0.33, 0.67, 1, 1.33, 1.67, 2, 2.33, 2.67, 3, 3.33, 3.67, 4, 4.50, 5, 6, 8, 10, 12, 14, 18 and 24 hours
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Albendazole IP 400 mg/ 400 mg - Test 1 (T1); Albendazole IP 400 mg/ 400 mg - Test 2 (T2); Albendazole 400 mg / IP 400mg- Reference 1 (R1); Albendazole 400 mg/ IP 400mg - Reference 2 (R2): Participants were orally administered with Albendazole (400 mg or 400 mg IP) tablet as single dose treatment under fed conditions on Day 1 in Periods 1, 2, 3 and 4
Arm/Group | Albendazole IP 400 mg/ 400 mg - Test 1 (T1) | Albendazole IP 400 mg/ 400 mg - Test 2 (T2) | Albendazole 400 mg / IP 400mg- Reference 1 (R1) | Albendazole 400 mg/ IP 400mg - Reference 2 (R2)
Number analyzed (Participants) | 63 | 60 | 63 | 62
ng*h/mL
  Albendazole | 189.347 (128.6) | 174.979 (119.0) | 169.433 (127.1) | 192.388 (116.1)
  Albendazole sulfoxide | 7372.856 (80.1) | 7189.644 (73.4) | 7204.107 (81.2) | 7816.474 (74.5)

6. Secondary Outcome: Time Until Cmax is Reached (Tmax) for Albendazole and Albendazole Sulfoxide
Description: as for outcome 5
Time Frame: Pre-dose, 0.33, 0.67, 1, 1.33, 1.67, 2, 2.33, 2.67, 3, 3.33, 3.67, 4, 4.50, 5, 6, 8, 10, 12, 14, 18 and 24 hours
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour (h)
Arm/Group | Albendazole IP 400 mg/ 400 mg - Test 1 (T1) | Albendazole IP 400 mg/ 400 mg - Test 2 (T2) | Albendazole 400 mg / IP 400mg- Reference 1 (R1) | Albendazole 400 mg/ IP 400mg - Reference 2 (R2)
Number analyzed (Participants) | 64 | 61 | 63 | 62
hour (h)
  Albendazole | 3.31 (33.4) | 3.41 (30.4) | 3.39 (32.9) | 3.52 (30.6)
  Albendazole sulfoxide | 4.64 (16.4) | 4.64 (21.7) | 4.62 (19.4) | 4.63 (20.0)

7. Secondary Outcome: Plasma Concentration Half-life (t1/2) of Albendazole and Albendazole Sulfoxide
Description: as for outcome 5
Time Frame: Pre-dose, 0.33, 0.67, 1, 1.33, 1.67, 2, 2.33, 2.67, 3, 3.33, 3.67, 4, 4.50, 5, 6, 8, 10, 12, 14, 18 and 24 hours
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour (h)
Arm/Group | Albendazole IP 400 mg/ 400mg - Test 1 (T1) | Albendazole IP 400 mg/ 400mg - Test 2 (T2) | Albendazole 400 mg/ IP 400mg - Reference 1 (R1) | Albendazole 400 mg/ IP 400mg - Reference 2 (R2)
Number analyzed (Participants) | 63 | 60 | 63 | 62
hour (h)
  Albendazole | 5.22 (55.1) | 5.53 (74.9) | 5.11 (60.0) | 5.62 (56.0)
  Albendazole sulfoxide | 8.47 (34.8) | 8.20 (28.4) | 8.21 (28.2) | 8.07 (32.8)

8. Secondary Outcome: Terminal Elimination Rate Constant (Lambda-z (λz)) of Albendazole and Albendazole Sulfoxide
Description: as for outcome 5
Time Frame: Pre-dose, 0.33, 0.67, 1, 1.33, 1.67, 2, 2.33, 2.67, 3, 3.33, 3.67, 4, 4.50, 5, 6, 8, 10, 12, 14, 18 and 24 hours
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/h
Arm/Group | Albendazole IP 400 mg/ 400 mg - Test 1 (T1) | Albendazole IP 400 mg/ 400mg - Test 2 (T2) | Albendazole 400 mg/ IP 400mg - Reference 1 (R1) | Albendazole 400 mg/ IP 400mg - Reference 2 (R2)
Number analyzed (Participants) | 63 | 60 | 63 | 62
1/h
  Albendazole | 0.133 (57.6) | 0.125 (61.8) | 0.136 (60.8) | 0.123 (43.8)
  Albendazole sulfoxide | 0.082 (29.3) | 0.085 (40.7) | 0.084 (33.0) | 0.086 (38.9)

9. Secondary Outcome: Observed Percentage of Extrapolated Area Under Concentration (AUC_% Extrap_obs) for Albendazole and Albendazole Sulfoxide
Description: as for outcome 5
Time Frame: Pre-dose, 0.33, 0.67, 1, 1.33, 1.67, 2, 2.33, 2.67, 3, 3.33, 3.67, 4, 4.50, 5, 6, 8, 10, 12, 14, 18 and 24 hours
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage
Groups:
- Albendazole IP 400 mg / 400mg- Test 1 (T1); Albendazole IP 400 mg/ 400mg - Test 2 (T2); Albendazole 400 mg/ IP 400mg - Reference 1 (R1); Albendazole 400 mg/ IP 400mg - Reference 2 (R2): Participants were orally administered with Albendazole (400 mg or 400 mg IP) tablet as single dose treatment under fed conditions on Day 1 in Periods 1, 2, 3 and 4
Arm/Group | Albendazole IP 400 mg / 400mg- Test 1 (T1) | Albendazole IP 400 mg/ 400mg - Test 2 (T2) | Albendazole 400 mg/ IP 400mg - Reference 1 (R1) | Albendazole 400 mg/ IP 400mg - Reference 2 (R2)
Number analyzed (Participants) | 63 | 63 | 60 | 62
Percentage
  Albendazole | 3.304 (111.2) | 3.241 (99.0) | 3.763 (112.6) | 3.275 (90.6)
  Albendazole sulfoxide | 14.513 (47.9) | 13.726 (45.7) | 13.795 (45.1) | 13.243 (50.8)

10. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: A TEAE is any event that was not present prior to the initiation of study treatment or any event already present that worsens in either intensity or frequency following exposure to study treatment.
Time Frame: Up to 22 days
Population: Safety Population included all randomized participants who received at least 1 dose of study medication. Each participant was counted once throughout the study for this analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Albendazole IP 400mg- Test (T): Participants received a single oral dose of 400 mg Albendazole Indian Pharmacopoeia (IP) tablet under fed conditions on Day 1 in either treatment Periods 1, 2, 3 and 4.
- Albendazole 400mg- Reference (R): Participants received a single oral dose of 400 mg Albendazole tablet under fed conditions on Day 1 in either treatment Periods 1, 2, 3 and 4.
Arm/Group | Albendazole IP 400mg- Test (T) | Albendazole 400mg- Reference (R)
Number analyzed (Participants) | 67 | 68
Participants | 7 | 6

11. Secondary Outcome: Absolute Values of Vital Signs: Blood Pressure (Diastolic and Systolic)
Description: Diastolic blood pressure (DBP) and systolic blood pressure (SBP) were collected in sitting position.
Time Frame: At pre-dose (within 60 minutes before the dosing) and at 2, 4, 6, 12 and 24 hours (Hrs) post-dose in each period
Population: Safety Population. As pre-specified in SAP, data for safety was collected and reported across two treatment groups as participants were randomized in either of the two treatment sequences (TRTR or RTRT) at the start of the study and they remained in the same sequence until end of the study. Each participant was counted once throughout the study for this analysis.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Groups:
- TRTR: Participants were orally administered with 400 milligram (mg) Albendazole Indian Pharmacopoeia (IP) - (T) tablet as single dose treatment under fed conditions on Day 1 in Period 1, followed by single dose treatment of 400 mg albendazole (R) tablets in Period 2, then 400 mg single dose of albendazole (T) further followed by 400 mg single dose of albendazole (R)
- RTRT: Participants were orally administered with 400 milligram (mg) Albendazole (R) tablet as single dose treatment under fed conditions on Day 1 in Period 1, followed by single dose treatment of 400 mg albendazole (T) tablets in Period 2, then 400 mg single dose of albendazole (R) further followed by 400 mg single dose of albendazole (T)
Arm/Group | TRTR | RTRT
Number analyzed (Participants) | 35 | 35
millimeters of mercury (mmHg)
  DBP - Period 1, Pre-dose | 76.1 (4.17) | 77.1 (4.32)
  DBP - Period 1, 2 Hrs Post Dose | 74.8 (3.47) | 75.7 (3.50)
  DBP - Period 1, 4 Hrs Post Dose | 74.6 (4.41) | 75.7 (4.29)
  DBP - Period 1, 6 Hrs Post Dose | 73.4 (5.20) | 71.4 (3.90)
  DBP - Period 1, 12 Hrs Post Dose | 73.9 (5.22) | 73.9 (4.70)
  DBP - Period 1, 24 Hrs Post Dose | 76.2 (3.71) | 75.5 (2.83)
  DBP - Period 2, Pre-Dose: number analyzed (Participants) | 31 | 31
  DBP - Period 2, Pre-Dose | 72.9 (3.26) | 75.7 (3.38)
  DBP - Period 2, 2 Hrs Post Dose: number analyzed (Participants) | 31 | 31
  DBP - Period 2, 2 Hrs Post Dose | 71.4 (5.55) | 71.9 (4.66)
  DBP - Period 2, 4 Hrs Post Dose: number analyzed (Participants) | 31 | 31
  DBP - Period 2, 4 Hrs Post Dose | 70.3 (4.13) | 71.5 (4.89)
  DBP - Period 2, 6 Hrs Post Dose: number analyzed (Participants) | 31 | 31
  DBP - Period 2, 6 Hrs Post Dose | 74.5 (2.29) | 74.2 (2.65)
  DBP - Period 2,12 Hrs Post Dose: number analyzed (Participants) | 31 | 31
  DBP - Period 2,12 Hrs Post Dose | 70.7 (5.62) | 73.2 (4.81)
  DBP - Period 2, 24 Hrs Post Dose: number analyzed (Participants) | 31 | 31
  DBP - Period 2, 24 Hrs Post Dose | 76.2 (3.52) | 76.7 (4.02)
  DBP - Period 3, Pre-Dose: number analyzed (Participants) | 32 | 32
  DBP - Period 3, Pre-Dose | 78.9 (3.17) | 78.9 (3.48)
  DBP - Period 3, 2 Hrs Post Dose: number analyzed (Participants) | 32 | 32
  DBP - Period 3, 2 Hrs Post Dose | 73.6 (5.56) | 75.1 (4.43)
  DBP - Period 3, 4 Hrs Post Dose: number analyzed (Participants) | 32 | 32
  DBP - Period 3, 4 Hrs Post Dose | 76.3 (5.47) | 73.3 (3.93)
  DBP - Period 3, 6 Hrs Post Dose: number analyzed (Participants) | 32 | 32
  DBP - Period 3, 6 Hrs Post Dose | 75.1 (6.18) | 74.4 (4.78)
  DBP - Period 3,12 Hrs Post Dose: number analyzed (Participants) | 32 | 32
  DBP - Period 3,12 Hrs Post Dose | 75.0 (4.49) | 73.4 (4.05)
  DBP - Period 3, 24 Hrs Post Dose: number analyzed (Participants) | 32 | 32
  DBP - Period 3, 24 Hrs Post Dose | 75.9 (2.80) | 75.7 (3.94)
  DBP - Period 4, Pre-Dose: number analyzed (Participants) | 31 | 30
  DBP - Period 4, Pre-Dose | 76.3 (3.47) | 76.0 (3.68)
  DBP - Period 4, 2 Hrs Post Dose: number analyzed (Participants) | 31 | 30
  DBP - Period 4, 2 Hrs Post Dose | 72.5 (4.79) | 73.7 (4.51)
  DBP - Period 4, 4 Hrs Post Dose: number analyzed (Participants) | 31 | 30
  DBP - Period 4, 4 Hrs Post Dose | 74.1 (2.61) | 73.8 (3.94)
  DBP - Period 4, 6 Hrs Post Dose: number analyzed (Participants) | 31 | 30
  DBP - Period 4, 6 Hrs Post Dose | 73.2 (2.86) | 73.8 (3.34)
  DBP - Period 4, 12 Hrs Post Dose: number analyzed (Participants) | 31 | 30
  DBP - Period 4, 12 Hrs Post Dose | 74.3 (3.47) | 74.7 (4.31)
  DBP - Period 4, 24 Hrs Post Dose: number analyzed (Participants) | 28 | 30
  DBP - Period 4, 24 Hrs Post Dose | 77.1 (2.46) | 75.6 (3.12)
  SBP - Period 1, Pre-dose | 116.1 (3.53) | 116.3 (3.22)
  SBP - Period 1, 2 Hrs Post Dose | 116.2 (3.46) | 116.9 (2.71)
  SBP - Period 1, 4 Hrs Post Dose | 116.3 (4.51) | 117.4 (3.99)
  SBP - Period 1, 6 Hrs Post Dose | 117.3 (4.60) | 119.5 (5.20)
  SBP - Period 1, 12 Hrs Post Dose | 116.5 (4.90) | 117.4 (4.02)
  SBP - Period 1, 24 Hrs Post Dose | 116.7 (3.29) | 117.0 (3.89)
  SBP - Period 2, Pre-dose: number analyzed (Participants) | 31 | 31
  SBP - Period 2, Pre-dose | 113.9 (4.50) | 116.4 (3.12)
  SBP - Period 2, 2 Hrs Post Dose: number analyzed (Participants) | 31 | 31
  SBP - Period 2, 2 Hrs Post Dose | 120.3 (4.64) | 119.8 (2.89)
  SBP - Period 2, 4 Hrs Post Dose: number analyzed (Participants) | 31 | 31
  SBP - Period 2, 4 Hrs Post Dose | 119.4 (2.55) | 120.3 (4.07)
  SBP - Period 2, 6 Hrs Post Dose: number analyzed (Participants) | 31 | 31
  SBP - Period 2, 6 Hrs Post Dose | 117.5 (3.90) | 116.8 (4.22)
  SBP - Period 2, 12 Hrs Post Dose: number analyzed (Participants) | 31 | 31
  SBP - Period 2, 12 Hrs Post Dose | 118.6 (4.45) | 119.6 (4.21)
  SBP - Period 2, 24 Hrs Post Dose: number analyzed (Participants) | 31 | 31
  SBP - Period 2, 24 Hrs Post Dose | 116.6 (3.70) | 117.0 (4.53)
  SBP - Period 3, Pre-dose: number analyzed (Participants) | 32 | 32
  SBP - Period 3, Pre-dose | 118.7 (3.12) | 117.9 (3.73)
  SBP - Period 3, 2 Hrs Post Dose: number analyzed (Participants) | 32 | 32
  SBP - Period 3, 2 Hrs Post Dose | 114.2 (4.14) | 115.7 (3.67)
  SBP - Period 3, 4 Hrs Post Dose: number analyzed (Participants) | 32 | 32
  SBP - Period 3, 4 Hrs Post Dose | 115.9 (3.88) | 114.8 (3.51)
  SBP - Period 3, 6 Hrs Post Dose: number analyzed (Participants) | 32 | 32
  SBP - Period 3, 6 Hrs Post Dose | 115.0 (4.40) | 115.2 (3.69)
  SBP - Period 3, 12 Hrs Post Dose: number analyzed (Participants) | 32 | 32
  SBP - Period 3, 12 Hrs Post Dose | 115.4 (3.39) | 115.1 (3.33)
  SBP - Period 3, 24 Hrs Post Dose: number analyzed (Participants) | 32 | 32
  SBP - Period 3, 24 Hrs Post Dose | 116.8 (3.89) | 116.0 (3.01)
  SBP - Period 4, Pre-dose: number analyzed (Participants) | 31 | 30
  SBP - Period 4, Pre-dose | 117.0 (3.18) | 116.4 (2.99)
  SBP - Period 4, 2 Hrs Post Dose: number analyzed (Participants) | 31 | 30
  SBP - Period 4, 2 Hrs Post Dose | 116.6 (3.20) | 116.3 (3.35)
  SBP - Period 4, 4 Hrs Post Dose: number analyzed (Participants) | 31 | 30
  SBP - Period 4, 4 Hrs Post Dose | 116.6 (3.91) | 115.9 (4.23)
  SBP - Period 4, 6 Hrs Post Dose: number analyzed (Participants) | 31 | 30
  SBP - Period 4, 6 Hrs Post Dose | 118.3 (3.43) | 119.1 (3.81)
  SBP - Period 4, 12 Hrs Post Dose: number analyzed (Participants) | 31 | 30
  SBP - Period 4, 12 Hrs Post Dose | 116.3 (3.69) | 115.6 (3.94)
  SBP - Period 4, 24 Hrs Post Dose: number analyzed (Participants) | 28 | 30
  SBP - Period 4, 24 Hrs Post Dose | 116.0 (3.13) | 115.2 (3.00)

12. Secondary Outcome: Absolute Values of Vital Signs: Respiratory Rate
Description: Respiratory rate was collected in sitting position.
Time Frame: At screening, after check-in and before check-out in each period (each period is of 1 day)
Population: Safety Population. As pre-specified in SAP, data for safety was collected and reported across two treatment groups as participants were randomized in either of the two treatment sequences (TRTR or RTRT) at the start of the study and they remained in the same sequence until end of the study. Each participant was counted once throughout the study for this analysis. Only those participants with data available in specified categories have been analyzed.
Measure: Mean (Standard Deviation); unit: breaths per minute (bpm)
Arm/Group | TRTR | RTRT
Number analyzed (Participants) | 35 | 35
breaths per minute (bpm)
  At Screening | 15.5 (2.08) | 15.8 (2.21)
  Period 1, after Check-in | 17.0 (2.13) | 16.4 (1.82)
  Period 1, before Check-out: number analyzed (Participants) | 33 | 34
  Period 1, before Check-out | 16.5 (2.69) | 16.5 (2.33)
  Period 2, after Check-in: number analyzed (Participants) | 32 | 33
  Period 2, after Check-in | 17.3 (2.72) | 16.8 (2.34)
  Period 2, before Check-out: number analyzed (Participants) | 32 | 33
  Period 2, before Check-out | 17.6 (2.41) | 16.8 (2.64)
  Period 3, after Check-in: number analyzed (Participants) | 33 | 32
  Period 3, after Check-in | 16.9 (2.24) | 17.6 (2.50)
  Period 3, before Check-out: number analyzed (Participants) | 33 | 32
  Period 3, before Check-out | 17.0 (1.95) | 16.3 (2.06)
  Period 4, after Check-in: number analyzed (Participants) | 31 | 31
  Period 4, after Check-in | 18.6 (2.20) | 18.3 (2.67)
  Period 4, before Check-out: number analyzed (Participants) | 28 | 31
  Period 4, before Check-out | 17.9 (2.28) | 17.7 (2.26)

13. Secondary Outcome: Absolute Values of Vital Signs: Radial Pulse
Description: Radial pulse was collected in sitting position.
Time Frame: At pre-dose (within 60 minutes before the dosing) and at 2, 4, 6, 12 and 24 hours post-dose in each period (each period is of 1 day)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | TRTR | RTRT
Number analyzed (Participants) | 35 | 35
beats per minute (bpm)
  Period 1, Pre-dose | 72.9 (6.31) | 74.2 (6.62)
  Period 1, 2 Hrs Post Dose | 70.6 (3.49) | 70.4 (3.39)
  Period 1, 4 Hrs Post Dose | 73.4 (4.38) | 72.9 (4.53)
  Period 1, 6 Hrs Post Dose | 72.8 (3.73) | 71.1 (4.37)
  Period 1, 12 Hrs Post Dose | 72.1 (4.80) | 70.7 (3.73)
  Period 1, 24 Hrs Post Dose | 72.7 (3.60) | 71.4 (3.68)
  Period 2, Pre-dose: number analyzed (Participants) | 31 | 31
  Period 2, Pre-dose | 72.4 (3.36) | 73.9 (5.48)
  Period 2, 2 Hrs Post Dose: number analyzed (Participants) | 31 | 31
  Period 2, 2 Hrs Post Dose | 67.4 (4.48) | 68.0 (4.20)
  Period 2, 4 Hrs Post Dose: number analyzed (Participants) | 31 | 31
  Period 2, 4 Hrs Post Dose | 67.9 (3.44) | 68.6 (4.20)
  Period 2, 6 Hrs Post Dose: number analyzed (Participants) | 31 | 31
  Period 2, 6 Hrs Post Dose | 72.8 (5.05) | 74.2 (4.39)
  Period 2, 12 Hrs Post Dose: number analyzed (Participants) | 31 | 31
  Period 2, 12 Hrs Post Dose | 70.2 (4.17) | 71.7 (5.41)
  Period 2, 24 Hrs Post Dose: number analyzed (Participants) | 31 | 31
  Period 2, 24 Hrs Post Dose | 69.2 (3.92) | 71.0 (3.26)
  Period 3, Pre-dose: number analyzed (Participants) | 32 | 32
  Period 3, Pre-dose | 75.6 (4.02) | 74.7 (6.32)
  Period 3, 2 Hrs Post Dose: number analyzed (Participants) | 32 | 32
  Period 3, 2 Hrs Post Dose | 69.6 (5.27) | 71.9 (3.95)
  Period 3, 4 Hrs Post Dose: number analyzed (Participants) | 32 | 32
  Period 3, 4 Hrs Post Dose | 70.8 (5.65) | 70.0 (3.66)
  Period 3, 6 Hrs Post Dose: number analyzed (Participants) | 32 | 32
  Period 3, 6 Hrs Post Dose | 70.7 (5.22) | 71.9 (4.38)
  Period 3, 12 Hrs Post Dose: number analyzed (Participants) | 32 | 32
  Period 3, 12 Hrs Post Dose | 73.0 (5.21) | 73.1 (3.52)
  Period 3, 24 Hrs Post Dose: number analyzed (Participants) | 32 | 32
  Period 3, 24 Hrs Post Dose | 70.9 (5.56) | 70.6 (4.05)
  Period 4, Pre-dose: number analyzed (Participants) | 31 | 30
  Period 4, Pre-dose | 75.0 (6.51) | 75.3 (7.10)
  Period 4, 2 Hrs Post Dose: number analyzed (Participants) | 31 | 30
  Period 4, 2 Hrs Post Dose | 69.6 (5.04) | 68.8 (3.99)
  Period 4, 4 Hrs Post Dose: number analyzed (Participants) | 31 | 30
  Period 4, 4 Hrs Post Dose | 72.2 (2.85) | 71.4 (4.17)
  Period 4, 6 Hrs Post Dose: number analyzed (Participants) | 31 | 30
  Period 4, 6 Hrs Post Dose | 72.2 (2.98) | 72.0 (2.52)
  Period 4, 12 Hrs Post Dose: number analyzed (Participants) | 31 | 30
  Period 4, 12 Hrs Post Dose | 70.6 (3.19) | 72.9 (3.10)
  Period 4, 24 Hrs Post Dose: number analyzed (Participants) | 28 | 30
  Period 4, 24 Hrs Post Dose | 69.9 (4.71) | 71.5 (5.20)

14. Secondary Outcome: Change From Baseline in Vital Signs: Blood Pressure
Description: Diastolic blood pressure (DBP) and systolic blood pressure (SBP) were collected in sitting position.
Time Frame: Pre-dose (within 60 minutes before the dosing) and at 2, 4, 6, 12 and 24 hours post-dose in each period
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | TRTR | RTRT
Number analyzed (Participants) | 35 | 35
millimeters of mercury (mmHg)
  DBP - Period 1, Pre-dose | 0.0 (0.00) | 0.0 (0.00)
  DBP - Period 1, 2 Hrs Post Dose | -1.3 (5.66) | -1.4 (5.71)
  DBP - Period 1, 4 Hrs Post Dose | -1.5 (6.44) | -1.4 (5.73)
  DBP - Period 1, 6 Hrs Post Dose | -2.7 (6.86) | -5.7 (6.14)
  DBP - Period 1, 12 Hrs Post Dose | -2.2 (7.29) | -3.2 (6.55)
  DBP - Period 1, 24 Hrs Post Dose | 0.1 (5.85) | -1.5 (4.60)
  DBP - Period 2, Pre-dose: number analyzed (Participants) | 31 | 31
  DBP - Period 2, Pre-dose | 0.0 (0.00) | 0.0 (0.00)
  DBP - Period 2, 2 Hrs Post Dose: number analyzed (Participants) | 31 | 31
  DBP - Period 2, 2 Hrs Post Dose | -1.5 (7.15) | -3.8 (5.57)
  DBP - Period 2, 4 Hrs Post Dose: number analyzed (Participants) | 31 | 31
  DBP - Period 2, 4 Hrs Post Dose | -2.6 (5.35) | -4.2 (6.23)
  DBP - Period 2, 6 Hrs Post Dose: number analyzed (Participants) | 31 | 31
  DBP - Period 2, 6 Hrs Post Dose | 1.5 (3.53) | -1.5 (4.06)
  DBP - Period 2, 12 Hrs Post Dose: number analyzed (Participants) | 31 | 31
  DBP - Period 2, 12 Hrs Post Dose | -2.2 (5.55) | -2.5 (5.70)
  DBP - Period 2, 24 Hrs Post Dose: number analyzed (Participants) | 31 | 31
  DBP - Period 2, 24 Hrs Post Dose | 3.3 (5.13) | 1.0 (5.93)
  DBP - Period 3, Pre-dose: number analyzed (Participants) | 32 | 32
  DBP - Period 3, Pre-dose | 0.0 (0.00) | 0.0 (0.00)
  DBP - Period 3, 2 Hrs Post Dose: number analyzed (Participants) | 32 | 32
  DBP - Period 3, 2 Hrs Post Dose | -5.3 (6.77) | -3.8 (5.09)
  DBP - Period 3, 4 Hrs Post Dose: number analyzed (Participants) | 32 | 32
  DBP - Period 3, 4 Hrs Post Dose | -2.6 (5.12) | -5.7 (4.37)
  DBP - Period 3, 6 Hrs Post Dose: number analyzed (Participants) | 32 | 32
  DBP - Period 3, 6 Hrs Post Dose | -3.8 (6.82) | -4.6 (6.18)
  DBP - Period 3, 12 Hrs Post Dose: number analyzed (Participants) | 32 | 32
  DBP - Period 3, 12 Hrs Post Dose | -3.9 (5.03) | -5.6 (5.15)
  DBP - Period 3, 24 Hrs Post Dose: number analyzed (Participants) | 32 | 32
  DBP - Period 3, 24 Hrs Post Dose | -2.9 (3.83) | -3.3 (4.89)
  DBP - Period 4, Pre-dose: number analyzed (Participants) | 31 | 30
  DBP - Period 4, Pre-dose | 0.0 (0.00) | 0.0 (0.00)
  DBP - Period 4, 2 Hrs Post Dose: number analyzed (Participants) | 31 | 30
  DBP - Period 4, 2 Hrs Post Dose | -3.8 (5.69) | -2.3 (4.60)
  DBP - Period 4, 4 Hrs Post Dose: number analyzed (Participants) | 31 | 30
  DBP - Period 4, 4 Hrs Post Dose | -2.3 (4.25) | -2.2 (5.24)
  DBP - Period 4, 6 Hrs Post Dose: number analyzed (Participants) | 31 | 30
  DBP - Period 4, 6 Hrs Post Dose | -3.1 (4.35) | -2.2 (4.34)
  DBP - Period 4, 12 Hrs Post Dose: number analyzed (Participants) | 31 | 30
  DBP - Period 4, 12 Hrs Post Dose | -2.0 (4.32) | -1.3 (5.62)
  DBP - Period 4, 24 Hrs Post Dose: number analyzed (Participants) | 28 | 30
  DBP - Period 4, 24 Hrs Post Dose | 0.6 (4.52) | -0.4 (4.38)
  SBP - Period 1, Pre-dose | 0.0 (0.00) | 0.0 (0.00)
  SBP - Period 1, 2 Hrs Post Dose | 0.1 (5.09) | 0.6 (4.10)
  SBP - Period 1, 4 Hrs Post Dose | 0.2 (5.50) | 1.1 (4.98)
  SBP - Period 1, 6 Hrs Post Dose | 1.1 (5.30) | 3.3 (6.21)
  SBP - Period 1, 12 Hrs Post Dose | 0.3 (5.69) | 1.1 (4.63)
  SBP - Period 1, 24 Hrs Post Dose | 0.6 (5.61) | 0.7 (5.72)
  SBP - Period 2, Pre-dose: number analyzed (Participants) | 31 | 31
  SBP - Period 2, Pre-dose | 0.0 (0.00) | 0.0 (0.00)
  SBP - Period 2, 2 Hrs Post Dose: number analyzed (Participants) | 31 | 31
  SBP - Period 2, 2 Hrs Post Dose | 6.4 (7.60) | 3.4 (3.39)
  SBP - Period 2, 4 Hrs Post Dose: number analyzed (Participants) | 31 | 31
  SBP - Period 2, 4 Hrs Post Dose | 5.5 (6.09) | 3.9 (5.35)
  SBP - Period 2, 6 Hrs Post Dose: number analyzed (Participants) | 31 | 31
  SBP - Period 2, 6 Hrs Post Dose | 3.6 (5.90) | 0.4 (5.12)
  SBP - Period 2, 12 Hrs Post Dose: number analyzed (Participants) | 31 | 31
  SBP - Period 2, 12 Hrs Post Dose | 4.8 (6.08) | 3.2 (4.64)
  SBP - Period 2, 24 Hrs Post Dose: number analyzed (Participants) | 31 | 31
  SBP - Period 2, 24 Hrs Post Dose | 2.8 (5.93) | 0.6 (6.10)
  SBP - Period 3, Pre-dose: number analyzed (Participants) | 32 | 32
  SBP - Period 3, Pre-dose | 0.0 (0.00) | 0.0 (0.00)
  SBP - Period 3, 2 Hrs Post Dose: number analyzed (Participants) | 32 | 32
  SBP - Period 3, 2 Hrs Post Dose | -4.5 (4.95) | -2.2 (4.58)
  SBP - Period 3, 4 Hrs Post Dose: number analyzed (Participants) | 32 | 32
  SBP - Period 3, 4 Hrs Post Dose | -2.8 (5.42) | -3.1 (4.98)
  SBP - Period 3, 6 Hrs Post Dose: number analyzed (Participants) | 32 | 32
  SBP - Period 3, 6 Hrs Post Dose | -3.7 (5.18) | -2.7 (4.84)
  SBP - Period 3, 12 Hrs Post Dose: number analyzed (Participants) | 32 | 32
  SBP - Period 3, 12 Hrs Post Dose | -3.3 (4.27) | -2.8 (5.32)
  SBP - Period 3, 24 Hrs Post Dose: number analyzed (Participants) | 32 | 32
  SBP - Period 3, 24 Hrs Post Dose | -1.9 (4.17) | -1.9 (4.13)
  SBP - Period 4, Pre-dose: number analyzed (Participants) | 31 | 30
  SBP - Period 4, Pre-dose | 0.0 (0.00) | 0.0 (0.00)
  SBP - Period 4, 2 Hrs Post Dose: number analyzed (Participants) | 31 | 30
  SBP - Period 4, 2 Hrs Post Dose | -0.4 (4.18) | -0.1 (3.82)
  SBP - Period 4, 4 Hrs Post Dose: number analyzed (Participants) | 31 | 30
  SBP - Period 4, 4 Hrs Post Dose | -0.4 (5.30) | -0.5 (4.67)
  SBP - Period 4, 6 Hrs Post Dose: number analyzed (Participants) | 31 | 30
  SBP - Period 4, 6 Hrs Post Dose | 1.3 (4.34) | 2.7 (3.66)
  SBP - Period 4, 12 Hrs Post Dose: number analyzed (Participants) | 31 | 30
  SBP - Period 4, 12 Hrs Post Dose | -0.7 (4.99) | -0.8 (5.67)
  SBP - Period 4, 24 Hrs Post Dose: number analyzed (Participants) | 28 | 30
  SBP - Period 4, 24 Hrs Post Dose | -0.9 (4.27) | -1.2 (3.66)

15. Secondary Outcome: Change From Baseline in Vital Signs: Respiratory Rate
Description: Respiratory rate was collected in sitting position.
Time Frame: After Check-in (Baseline) and before Check-out for each period (each period is of 1 day)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: breaths per minute (bpm)
Arm/Group | TRTR | RTRT
Number analyzed (Participants) | 33 | 34
breaths per minute (bpm)
  Period 1 | -0.6 (3.72) | 0.2 (2.26)
  Period 2: number analyzed (Participants) | 32 | 33
  Period 2 | 0.6 (3.56) | 0.4 (3.91)
  Period 3: number analyzed (Participants) | 33 | 32
  Period 3 | 0.2 (2.53) | -0.0 (3.27)
  Period 4: number analyzed (Participants) | 28 | 31
  Period 4 | 0.9 (3.41) | 1.3 (3.07)

16. Secondary Outcome: Change From Baseline in Vital Signs: Radial Pulse
Description: Radial pulse was collected in sitting position.
Time Frame: pre-dose (within 60 minutes before the dosing) and at 2, 4, 6, 12 and 24 hours post-dose in each period
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | TRTR | RTRT
Number analyzed (Participants) | 35 | 35
beats per minute (bpm)
  Period 1, Pre-dose | 0.0 (0.00) | 0.0 (0.00)
  Period 1, 2 Hrs Post Dose | -2.2 (6.86) | -3.8 (7.79)
  Period 1, 4 Hrs Post Dose | 0.6 (7.57) | -1.3 (9.23)
  Period 1, 6 Hrs Post Dose | -0.1 (7.87) | -3.0 (7.71)
  Period 1, 12 Hrs Post Dose | -0.7 (8.85) | -3.4 (7.89)
  Period 1, 24 Hrs Post Dose | -0.1 (7.64) | -2.7 (7.96)
  Period 2, Pre-dose: number analyzed (Participants) | 31 | 31
  Period 2, Pre-dose | 0.0 (0.00) | 0.0 (0.00)
  Period 2, 2 Hrs Post Dose: number analyzed (Participants) | 31 | 31
  Period 2, 2 Hrs Post Dose | -5.0 (5.08) | -5.9 (5.40)
  Period 2, 4 Hrs Post Dose: number analyzed (Participants) | 31 | 31
  Period 2, 4 Hrs Post Dose | -4.5 (5.05) | -5.4 (6.23)
  Period 2, 6 Hrs Post Dose: number analyzed (Participants) | 31 | 31
  Period 2, 6 Hrs Post Dose | 0.5 (5.95) | 0.3 (6.98)
  Period 2, 12 Hrs Post Dose: number analyzed (Participants) | 31 | 31
  Period 2, 12 Hrs Post Dose | -2.2 (5.71) | -2.2 (8.41)
  Period 2, 24 Hrs Post Dose: number analyzed (Participants) | 31 | 31
  Period 2, 24 Hrs Post Dose | -3.2 (5.58) | -2.9 (6.47)
  Period 3, Pre-dose: number analyzed (Participants) | 32 | 32
  Period 3, Pre-dose | 0.0 (0.00) | 0.0 (0.00)
  Period 3, 2 Hrs Post Dose: number analyzed (Participants) | 32 | 32
  Period 3, 2 Hrs Post Dose | -6.0 (6.41) | -2.8 (6.70)
  Period 3, 4 Hrs Post Dose: number analyzed (Participants) | 32 | 32
  Period 3, 4 Hrs Post Dose | -4.8 (5.47) | -4.7 (7.09)
  Period 3, 6 Hrs Post Dose: number analyzed (Participants) | 32 | 32
  Period 3, 6 Hrs Post Dose | -4.9 (6.32) | -2.8 (7.72)
  Period 3, 12 Hrs Post Dose3: number analyzed (Participants) | 32 | 32
  Period 3, 12 Hrs Post Dose3 | -2.6 (7.82) | -1.6 (7.07)
  Period 3, 24 Hrs Post Dose: number analyzed (Participants) | 32 | 32
  Period 3, 24 Hrs Post Dose | -4.7 (6.73) | -4.1 (7.71)
  Period 4, Pre-dose: number analyzed (Participants) | 31 | 30
  Period 4, Pre-dose | 0.0 (0.00) | 0.0 (0.00)
  Period 4, 2 Hrs Post Dose: number analyzed (Participants) | 31 | 30
  Period 4, 2 Hrs Post Dose | -5.4 (8.94) | -6.5 (8.23)
  Period 4, 4 Hrs Post Dose: number analyzed (Participants) | 31 | 30
  Period 4, 4 Hrs Post Dose | -2.8 (8.16) | -3.9 (8.44)
  Period 4, 6 Hrs Post Dose: number analyzed (Participants) | 31 | 30
  Period 4, 6 Hrs Post Dose | -2.8 (7.09) | -3.3 (6.53)
  Period 4, 12 Hrs Post Dose: number analyzed (Participants) | 31 | 30
  Period 4, 12 Hrs Post Dose | -4.4 (7.27) | -2.3 (7.30)
  Period 4, 24 Hrs Post Dose: number analyzed (Participants) | 28 | 30
  Period 4, 24 Hrs Post Dose | -5.1 (7.73) | -3.8 (8.34)

ADVERSE EVENTS:
Time Frame: All cause mortality, non-serious adverse events (Non-SAEs) and serious adverse events (SAEs) were collected through the entire study duration of up to a maximum of 22 days.
Description: Safety Population included all randomized participants who received at least 1 dose of study medication. Each participant was counted once throughout the study for this analysis.
Arm/Group | Albendazole IP 400mg- Test (T) | Albendazole 400mg- Reference (R)
All-Cause Mortality (participants affected / at risk) | 0/67 | 0/68
Serious Adverse Events (participants affected / at risk) | 1/67 | 0/68
Other Adverse Events (participants affected / at risk) | 6/67 | 6/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Albendazole IP 400mg- Test (T) (N=67) | Albendazole 400mg- Reference (R) (N=68)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Albendazole IP 400mg- Test (T) (N=67) | Albendazole 400mg- Reference (R) (N=68)
Asthenia (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 3 (3)
Nasopharyngitis (Infections and infestations) | 2 (2) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (2) | 2 (3)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-07-04): https://cdn.clinicaltrials.gov/large-docs/59/NCT06201559/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-04): https://cdn.clinicaltrials.gov/large-docs/59/NCT06201559/SAP_001.pdf